CLINICAL TRIAL: NCT03048799
Title: Radiofrequency in the Treatment of Urinary Incontinence After Radical Prostatectomy: Randomized Clinical Trial
Brief Title: Radiofrequency in the Treatment of Urinary Incontinence After Radical Prostatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro de Atenção ao Assoalho Pélvico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U1111-1192-4467
Record Dates: First submitted 2017-02-02; First posted 2017-02-09 (Estimated); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Urinary Incontinence; Post Prostatectomy
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency on and Kinesiotherapy (Active Comparator): The radiofrequency application protocol with CAPENERGY device, which has two electrodes: an active one, which will be introduced into the anal region, using a condom and gel to The emission of radiofrequency and another electrode, dispersive, coupled to the patient's hip, which will function as earth. The temperature used in the treatment will be 41 ° C, which this parameter will be placed in the equipment, maintained for 2 minutes. Five RF sessions will be performed, with a seven-day interval between them. For the application, participants will be placed in lateral decubitus position. The session will be quick, with an average duration of 20 minutes.Kinesiotherapy will be done once a week, totaling five sessions. Initially, verbal information about location, function, and the correct way to contract the pelvic floor (PA) will be given.
  Interventions: Device: Radiofrequency
- Radiofrequency off and Kinesiotherapy (Placebo Comparator): The patient will be in lateral decubitus, the anal probe of the radiofrequency apparatus will be introduced, with the gel previously heated. The radio frequency will be off.
  Kinesiotherapy will be done once a week, totaling five sessions. Initially, verbal information about location, function, and the correct way to contract the pelvic floor (PA) will be given. In addition, at this point will be advised on the performance of "The Knack", which is a pre-contraction of the PA during the performance of some abdominal effort such as coughing, sneezing or laughing.
  Interventions: Device: Radiofrequency

INTERVENTIONS:
Device: Radiofrequency — The radiofrequency application protocol will be used in the form of capacitive electrical transfer, bipolar configuration, with CAPENERGY device (Figure 1), which has two electrodes: an active one, which will be introduced into the anal region, using a condom and gel to The emission of radiofrequency and another electrode, dispersive, coupled to the patient's hip, which will function as earth. The active electrode has at its end a sensor capable of capturing the temperature. The temperature used in the treatment will be 41 ° C, which this parameter will be placed in the equipment. Upon reaching the desired heating, the apparatus maintains the temperature and thus the application of the radiofrequency will be maintained for 2 minutes.

SUMMARY:
Post-prostatectomy urinary incontinence (IUPP) is a difficult to treat complication that causes a profound negative impact on the individual's quality of life, as well as seriously disrupts the physician-patient relationship and is a substantial public health problem . Urinary incontinence (UI) can occur both in the treatment of benign prostatic hyperplasia (BPH) and in the treatment of prostate cancer.

In the treatment of benign disease, this complication is associated with a very low prevalence, initially of 9% and about 1% in 12 months postoperatively. In radical prostatectomy, the prevalence is higher, varying from 2% to 87%, depending on the populations and sites studied, the definitions used, the different methodologies employed in the evaluation of incontinence, and also the different degrees of intensity of the disease . Several authors have evaluated the incidence of incontinence after robotic radical prostatectomy, open and laparoscopically. With these techniques, the reported total UI incidence varies from 4% to 40% .

With the high prevalence of IUPP, accelerating the recovery of urinary control is an important priority for patients and their caregivers, and the search for effective and low-risk treatments is a constant. Thus, the possibility of treatment with the radiofrequency (RF) feature arises.

DETAILED DESCRIPTION:
A current treatment proposal is the use of radiofrequency, which is a diathermic process generated by the radiation of an electromagnetic spectrum, resulting in an immediate retraction of existing collagen and subsequent activation of fibroblasts causing a neocollagenesis. In studies using radiofrequency to treat SUI, a therapeutic response to 50% was shown. Representing a more cost-effective treatment than surgery.

ELIGIBILITY:
Inclusion Criteria:

* will be individuals from 18 to 65 years of age with clinical complaints of urinary incontinence after prostatectomy and who agree to voluntarily participate in the research.

Exclusion Criteria:

* Will be excluded from the study the patients with time less than 45 days postoperative, difficulty understanding the proposed instruments, patients with neurological degenerative chronic diseases, patients with implantable cardioverter defibrillators and carriers of iatrogenic metals in the pelvic region.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2016-12-05 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2024-12-05 (Estimated)

PRIMARY OUTCOMES:
Pad Test (grams) | 1 month
  The pad test aims to quantify the urinary loss in different physical activities in the period of 1 hour.

SECONDARY OUTCOMES:
Pad Test (grams) | 6 month after
  The pad test aims to quantify the urinary loss in different physical activities in the period of 1 hour.
Quality of life Scale Questionaire | 1 month after
  Scale questionaire
Quality of life Scale Questionaire | 6 month after
  Scale questionaire
Quality of life Scale Questionaire | 1 year after
  Scale questionaire
Erectile dysfunction | 1 month
  A questionnaire with 15 questions will be applied in which it evaluates the erectile dysfunction, the name of questionnaire is International Index of Erectile Dysfunction (IIEF-5)
Erectile dysfunction | 6 month
  A questionnaire with 15 questions will be applied in which it evaluates the erectile dysfunction, the name of questionnaire is International Index of Erectile Dysfunction (IIEF-5)
quality of life specified urinary incontinence | 1 month
  The ICIQ-SF is a self-administered questionnaire composed of four questions that assess the frequency, severity and impact of UI, as well as a set of eight self-diagnosis items related to the causes or UI situations experienced by the respondents. The final score is found from the sum of the score of questions 3, 4 and 5. The overall score ranges from 0 to 21 points and the higher the score the greater the impact on the quality of life. The impact on the quality of life is divided in such a way: no impact (0 point); Light impact (from 1 to 3 points); Moderate impact (from 4 to 6 points); Serious impact (from 7 to 9 points); And very serious impact (10 or more points
quality of life specified urinary incontinence | 6 month
  The ICIQ-SF is a self-administered questionnaire composed of four questions that assess the frequency, severity and impact of UI, as well as a set of eight self-diagnosis items related to the causes or UI situations experienced by the respondents. The final score is found from the sum of the score of questions 3, 4 and 5. The overall score ranges from 0 to 21 points and the higher the score the greater the impact on the quality of life. The impact on the quality of life is divided in such a way: no impact (0 point); Light impact (from 1 to 3 points); Moderate impact (from 4 to 6 points); Serious impact (from 7 to 9 points); And very serious impact (10 or more points

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Atenção ao assoalho pélvico, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No